CLINICAL TRIAL: NCT05666453
Title: A Multi-center, Prospective, Randomized, Controlled, Open-label, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of Intravenous Immunoglobulin to Prevent Biliary Complications After ABO Incompatible Adult to Adult Living Donor Liver Transplantation
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of LIV-GAMMA SN Inj. in ABO-Incompatible Liver Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change of Clincal Development Plan
Sponsor: SK Plasma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SK_LIV_ABO
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment group (Experimental): LIV-GAMMA SN Inj. administration after ABO-incompatible liver transplantation
  Interventions: Biological: LIV-GAMMA SN Inj.
- Comparator group (Other): No administration after ABO-incompatible liver transplantation
  Interventions: Other: No intervention
- Reference group (Other): No administration after ABO-compatible liver transplantation
  Interventions: Other: No intervention

INTERVENTIONS:
Biological: LIV-GAMMA SN Inj. — LIV-GAMMA SN Inj. is administered at a dose of 0.6 g/kg/day from anhepatic phase to Day 2 post-operative to patients undergoing ABO-incompatible liver transplantation as an experimental group.
  Arms: Treatment group
Other: No intervention — None of investigational drugs are administered to patients.
  Arms: Comparator group; Reference group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of LIV-GAMMA SN Inj. administered for consecutive 3 days in adult subjects to prevent biliary complications after ABO incompatible adult to adult living donor liver transplantation (LDLT). The primary objective of this study is to determine the incidence rate of biliary complications for 48 weeks after liver transplantation. Incidence rate of transplant rejection, DSA, antibody reaction, CMV infection, infectious complications, DIHBS and recurrence rate of HCC as well as adverse events are assessed as additional efficacy and safety endpoints in this study.

ELIGIBILITY:
Inclusion Criteria:

* Completed informed consent process
* Male or female aged ≥19 years and <75 years
* Patients scheduled hospitalization for liver transplantation

Exclusion Criteria:

* Patients who are scheduled or have history of re-transplantation or multiorgan transplantation
* Patients receiving living donor in emergency
* Patients with Donor Specific Antibody (DSA) ≥ MFI 10,000 or Human Leukocyte Antigen (HLA) crossmatch (+) cytotoxic T-cell ≥ 1:32
* Patients with a history of biliary tract disease
* Patients who plasma exchange is forbidden (with a history of allergic or anaphylactic reaction to FFP, albumin, heparin, etc.)
* Patients with a history of specific medical conditions

  * Severe renal failure (eGFR < 30 mL/min/1.73 m^2 at screening)
  * Deep Vein Thrombosis (DVT) or thrombotic complications from Intravenous Immunoglobulin (IVIg) therapy
  * Cerebrovascular or cardiovascular disease (Hyperviscosity syndrome, Transient Ischemic Attack (TIA), Stroke, Thromboembolism, Unstable angina, etc.)
  * Clinical state causing secondary immunodeficiency (Leukemia, Lymphoma, Multiple myeloma, HIV infection, Chronic or Cyclic neutropenia (Absolute neutrophil < 500/mm^3), etc.)
  * Uncontrolled hypertension (Systolic blood pressure > 160 mmHg or Diastolic blood pressure > 100 mmHg)
  * Hemolytic or hemorrhagic anemia
  * Decreased cardiac functions
  * Bacterial, fungal or viral infection making liver transplantation forbidden
* Intraductal or vascular infiltration observed in patients with hepatocellular carcinoma using medical imaging before liver transplantation
* Patients metastasized to organs except for liver or diagnosed cancer except for liver cancer and squamous cell carcinoma within 5 years from screening
* Patients with sepsis
* Patients who had interventional therapy in blood vessels (hepatic vein, portal vein, hepatic artery, etc.) or bile ducts before LDLT
* Patients who have allergy or hypersensitivity to blood products, blood-derived products, IVIg or immunoglobulin G (IgG) products
* Patients who have immunoglobulin A (IgA) deficiency or anti-IgA antibody
* Patients who are pregnant and nursing
* Patients unwilling to use adequate method of contraception (hormonal methods, intrauterine device or intrauterine system, vasectomy, tubal ligation, etc.) during this study
* Patients who had received other investigational products within 8 weeks from complete consent or who are scheduled to receive other investigational products during this study
* Others whom the investigator considers ineligible for the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of biliary complications | 48 weeks
  The number and rate of subjects with biliary complications including cholangitis, biliary leaks or biliary strictures for 48 weeks after liver transplantation (Experimental group vs. Comparator group)

SECONDARY OUTCOMES:
Rate of transplant rejection | 48 weeks
  The number and rate of subjects with transplant rejection for 48 weeks after liver transplantation
Rate of Donor Specific Antibody (DSA) | 48 weeks
  The number and rate of subjects with Donor Specific Antibody (DSA) for 48 weeks after liver transplantation
Rate of antibody reaction by ABO subtype | 48 weeks
  The number and rate of subjects with antibody reaction by ABO subtype analysis for 48 weeks after liver transplantation
Rate of Cytomegalovirus (CMV) infection | 48 weeks
  The number and rate of subjects with Cytomegalovirus (CMV) infection for 48 weeks after liver transplantation
Rate of infectious complications | 48 weeks
  The number and rate of subjects with infectious complications for 48 weeks after liver transplantation
Rate of Diffuse Intrahepatic Biliary Stricture (DIHBS) | 48 weeks
  The number and rate of subjects with Diffuse Intrahepatic Biliary Stricture (DIHBS) for 48 weeks after liver transplantation
Recurrence rate of Hepatocellular Carcinoma (HCC) | 48 weeks
  The recurrence rate of subjects with Hepatocellular Carcinoma (HCC) for 48 weeks after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Joon Yi, MD, Study Chair — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam
  - Chung-Ang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul